CLINICAL TRIAL: NCT02506647
Title: A Phase 1, Exploratory, Randomized, Double-Blind, Two-Way Cross Over Study to Assess Pharmacokinetic and Pharmacodynamic Effects of Gan & Lee's Insulin Glargine Injection in Comparison to Lantus in Subjects With Type 1 Diabetes Mellitus
Brief Title: PK/PD Study of Gan & Lee's Insulin Glargine Injection in Comparison to Lantus in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GL-GLA-001
Record Dates: First submitted 2015-07-16; First posted 2015-07-23 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gallium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Gan & Lee insulin glargine followed by Lantus
  Interventions: Drug: Gan & Lee insulin glargine followed by Lantus
- Sequence 2 (Active Comparator): Lantus followed by Gan & Lee insulin glargine
  Interventions: Drug: Lantus followed by Gan & Lee insulin glargine

INTERVENTIONS:
Drug: Gan & Lee insulin glargine followed by Lantus — 0.4 IU/kg Gan & Lee insulin glargine injection SC, Lantus 0.4 IU/kg injection SC
  Arms: Sequence 1
Drug: Lantus followed by Gan & Lee insulin glargine — Lantus 0.4 IU/kg injection SC, 0.4 IU/kg Gan & Lee insulin glargine injection SC,
  Arms: Sequence 2

SUMMARY:
This is a Phase 1, exploratory, single dose, randomized, double-blind, two-way cross over, pilot, glucose clamp study to assess pharmacokinetic and pharmacodynamic effects of Gan & Lee's insulin glargine injection in comparison to the marketed Lantus (US) in subjects with type 1 diabetes mellitus (T1DM).

ELIGIBILITY:
Inclusion Criteria:

1. Female and Male subjects with T1DM, duration ≥12 months.
2. Adults ≥ 18 to ≤ 65 years of age.
3. Body mass index (BMI) ≥ 18.5 to ≤ 30.0 kg/m2.
4. Weight ≥ 50 kg.
5. Fasting serum C-peptide ≤ 0.4 nmol/L, assessed at a plasma glucose concentration > 90mg/dL.
6. HbA1c ≤ 9.5%.
7. Current stable treatment with insulin (consistent therapy with multiple daily injections with basal and bolus insulin or CSII).
8. Current stable dose of insulin (± 20% difference in total daily insulin dose) over the 2-week period prior to screening; total daily dose ≤ 1.2 IU/kg.
9. Female subjects must be non-pregnant and non-lactating. For postmenopausal females (no menses >12 months); postmenopausal status will be confirmed through testing of FSH levels ≥ 40 IU/mL at screening for subjects <55 years of age.
10. Ability to provide written informed consent.

Exclusion Criteria:

1. A subject who has proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
2. History of ≥ 2 episodes of severe hypoglycemia (as defined per ADA criteria) or ≥ 1 episodes of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within 6 months prior to screening.
3. Subjects is on a carbohydrate restricted diet (i.e., a diet < 100 grams per day of carbohydrate).
4. Systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 95 mmHg at screening. Treatment with no more than 2 antihypertensive medications must be with stable doses for at least 3 months prior to screening.
5. Current use of any drugs (other than insulin) that are known to interfere with glucose or insulin metabolism, including but not limited to oral corticosteroids, monoamino oxidase (MAO) inhibitors, growth hormone and non-selective β-blockers, loop diuretics.
6. Thyroid hormone use not stable during the past 3 months prior to dosing.
7. Hyperlipidemia treatment not on stable dose for ≥ 3 months prior to dosing. (HMG-CoA reductase inhibitor (statin), a fibrate (i.e. fenofibrate, gemfibrozil) and ezetimibe are allowed as treatment).
8. Any use of non-steroid anti-inflammatory drugs (NSAIDs) except for low-dose Aspirin is not allowed within 7 days prior to dosing and on the dosing day.
9. Participation in an investigational study within 30 days prior to dosing or 5 half-lives within the last dose of investigational product whichever is longer.
10. History of any major surgery within 6 months prior to screening.
11. History of any serious adverse reaction or hypersensitivity to insulin, insulin analogue, any of the product components, or chemically related products.
12. History of renal disease or abnormal kidney function tests at screening (glomerular filtration rate (GFR) < 60 mL/min/1.73m2 ).
13. Clinically significant abnormal hematology or biochemistry screening tests.
14. Any history of heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, coronary artery bypass graft surgery, or angioplasty, unstable angina requiring medication, transient ischemic attack, cerebral infarct, or cerebral hemorrhage.
15. History of any clinically significant gastrointestinal, cardiovascular, hematological, psychiatric, renal, hepatic, pancreatic or neurological abnormality as judged by the Investigator.
16. Personal or family history of hypercoagulability or thromboembolic disease.
17. History of any active infection, other than mild or viral illness within 30 days prior to dosing as judged by the Investigator.
18. History of alcohol or illicit/recreational drug abuse as judged by the Investigator within approximately 1 year. (Use of up to 1000 mL beer, 500 mL wine, or 100 mL distilled spirits is allowed).
19. Smoking > 10 cigarettes or equivalent use of any tobacco product (e.g.nicotine patch) within 6 months prior to Screening. Subjects must be able to refrain from smoking at least 1 week prior to admission and during each in-house period.
20. Known history of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibody.
21. Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution or metabolism of the drugs or the tolerability/safety measurements.
22. Presence of clinically significant physical, laboratory, or electrocardiogram (ECG) findings (e.g., QTcF > 470 msec for females, > 450 msec for males, LBBB) at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results.
23. Donation or loss of > 500 mL of blood or blood product within 56 days of dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effects | 0-24 hours
  Pharmacodynamic effects: Area under the glucose infusion rate, AUC GIR(0-24hr)
Pharmacokinetic effects | 0-24 hours
  Area under the insulin concentration-time curve, AUCINS (0-24hr)

SECONDARY OUTCOMES:
Pharmacokinetic effects | 0-12 hours
  AUCINS (0-12hr)
Pharmacokinetic effects | 12-24 hours
  AUCINS (12-24hr)
Pharmacodynamic effects | 0-12hours
  AUCGIR (0-12hr)
Pharmacodynamic effects | 12-24 hours
  AUCGIR (12-24hr)
Safety assessment as measured by incidence and severity of adverse events | 0-24 hours
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, San Diego, California, United States